CLINICAL TRIAL: NCT05899777
Title: Research, Development and Promotion of the Service Package of Yizhi Baduanjin for Mild Cognitive Impairment
Brief Title: Intervention Effect of Yizhi Baduanjin on Patients With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZY(2021-2023)-0105-B99
Record Dates: First submitted 2023-04-17; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Baduanjin
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): After proficiently mastering the complete set of Yizhi Baduanjin, the practice group is required to practice sitting posture of YizhiBaduanjin twice a day and standing posture of YizhiBaduanjin once every two days.
  Interventions: Other: Yizhi Baduanjin
- control group (No Intervention): The control group is a waiting control group, and after 24 weeks, they will continue to learn the Yizhi Baduanjin.

INTERVENTIONS:
Other: Yizhi Baduanjin — Yizhi Baduanjin is a newly compiled routine developed on the foundation of the traditional Baduanjin, aiming at the mental and cerebral health of middle-aged and elderly population, which combining the preliminary research result and principles of the traditional routine. It could be practiced in long term to prevent MCI and AD, or simply as a general health exercise for elders.
  Arms: Treatment group

SUMMARY:
With mild cognitive impairment (MCI) as the research object, the intervention effect of Yizhi Baduanjin on mild cognitive impairment was evaluated by using the Montreal Cognitive Assessment (MoCA) scale, human-computer interactive electronic cognitive function score, multi-measure EEG data and other evaluation indicators, with the intervention measures of Yizhi Baduanjin created by the Tai Chi Health Center in the early stage. This project is based on the preliminary study, followed the principles and methods of clinical epidemiology and evidence-based medicine, and designed a prospective, randomized, single-blind, parallel controlled trial to make up for the deficiency of existing drugs in the intervention of mild cognitive impairment, and to provide evidence for the clinical and community promotion and application of effective and safe traditional Chinese medicine non-pharmaceuticals in the prevention and treatment of mild cognitive impairment.

DETAILED DESCRIPTION:
Mild cognitive impairment（MCI） is a critical state between normal aging and dementia, with its core symptom being age-related cognitive decline. This critical state provides a window of opportunity for preventing Alzheimer's disease. At present, there is a lack of sufficient intervention methods to improve MCI.

Yizhi Baduanjin is an adaptation of traditional Baduanjin, which is more suitable for middle-aged and elderly people to practice and optimize for improving cognitive function. Previous observations and studies have provided some evidence to prove the beneficial effect of Yizhi Baduanjin on MCI.

This is a two-group prospective, randomized, assessor-blinded trial, planning to enroll 100 participants.They will randomly divided into two groups: the training group with 50 cases and the control group with 50 cases. The training group will receive intervention with the Yizhi Baduanjin, and various evaluation indicators will test before and 4、12、24 weeks after the intervention. The control group is a waiting control group, and after 24 weeks, they will continue to learn the Yizhi Baduanjin. The control group and the practice group will be tested simultaneously at four time points. Finally, the intervention effect will be evaluated through inter group and intra group comparisons of test data.

The main research purpose is to evaluate the clinical effect of Yizhi Baduanjin on MCI.The secondary research objective is to explore the possible mechanism of Yizhi Baduanjin in improving MCI.

ELIGIBILITY:
Inclusion Criteria:

* Subjective symptoms include memory loss
* MoCA score is less than 26 points
* No disability, no communication barrier, and can complete the cognitive function test of human-computer interaction
* Agree to participate in the project and sign the informed consent form

Exclusion Criteria:

* Alzheimer's patients
* Cognitive impairment caused by depression, cerebrovascular accident and other specific reasons
* Those who are unwilling or unable to take part in the Yizhi Baduanjin exercise

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
MoCA | Change from Baseline MOCA at 4 weeks
  The MoCA (Montreal Cognitive Assessment) is a tool used to assess cognitive function, primarily for the early detection of mild cognitive impairment and dementia.
  The MoCA scale consists of 30 questions, including evaluations of memory, attention, language, abstraction, orientation, spatial ability, and executive function. The scale includes more specific testing items, such as clock-drawing, reaction time, and number string recall. Each question has a standard answer or scoring criteria, and scores are totaled to a maximum of 30 points.The cutoffs for MCI are <26.
MoCA | Change from 4 weeks MOCA at 12 weeks
  The MoCA (Montreal Cognitive Assessment) is a tool used to assess cognitive function, primarily for the early detection of mild cognitive impairment and dementia.
  The MoCA scale consists of 30 questions, including evaluations of memory, attention, language, abstraction, orientation, spatial ability, and executive function. The scale includes more specific testing items, such as clock-drawing, reaction time, and number string recall. Each question has a standard answer or scoring criteria, and scores are totaled to a maximum of 30 points.The cutoffs for MCI are <26.
MoCA | Change from 12 weeks MOCA at 24 weeks
  The MoCA (Montreal Cognitive Assessment) is a tool used to assess cognitive function, primarily for the early detection of mild cognitive impairment and dementia.
  The MoCA scale consists of 30 questions, including evaluations of memory, attention, language, abstraction, orientation, spatial ability, and executive function. The scale includes more specific testing items, such as clock-drawing, reaction time, and number string recall. Each question has a standard answer or scoring criteria, and scores are totaled to a maximum of 30 points.The cutoffs for MCI are <26.

SECONDARY OUTCOMES:
Cognitive Function Score | Change from Baseline cognitive function score at 4 weeks
  Objective scores for the four cognitive tasks of "positional circle", "numerical circle", "numerical string", and "operation" in the MCI screening tool.
Cognitive Function Score | Change from 4 weeks cognitive function score at 12 weeks
  Objective scores for the four cognitive tasks of "positional circle", "numerical circle", "numerical string", and "operation" in the MCI screening tool.
Cognitive Function Score | Change from 12 weeks cognitive function score at 24 weeks
  Objective scores for the four cognitive tasks of "positional circle", "numerical circle", "numerical string", and "operation" in the MCI screening tool.
EEG data | Change from Baseline EEG data at 4 weeks
  EEG power spectrum, ApEn approximate entropy, LZ complexity, RE, NR correlation
EEG data | Change from 4 weeks EEG data at 12 weeks
  EEG power spectrum, ApEn approximate entropy, LZ complexity, RE, NR correlation
EEG data | Change from 12 weeks EEG data at 24 weeks
  EEG power spectrum, ApEn approximate entropy, LZ complexity, RE, NR correlation

IPD SHARING:
Plan to Share IPD: No